CLINICAL TRIAL: NCT00245154
Title: A Phase II/III Double Blind Randomized Trial of AZD2171 Versus Placebo in Patients Receiving Paclitaxel/Carboplatin Chemotherapy for the Treatment of Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Paclitaxel + Carboplatin With/Out Cediranib Maleate in Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR24; CAN-NCIC-BR24 (Other: PDQ); ZENECA-CAN-NCIC-BR24 (Other: Zeneca Group); FHCRC-6107 (Other: Search Results Web result with site links Fred Hutchinson Cancer Research Center); UWCC-UW 6107; UWCC- 06-2707-H/B; CDR0000450850 (Other: PDQ)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; cediranib; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral cediranib maleate once daily in the absence of disease progression or unacceptable toxicity. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment with paclitaxel and carboplatin repeats every 21 days for 6-8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: carboplatin; Drug: cediranib maleate; Drug: paclitaxel
- Arm II (Active Comparator): Patients receive oral placebo once daily in the absence of disease progression or unacceptable toxicity. Patients also receive paclitaxel and carboplatin as in arm I.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Other: placebo

INTERVENTIONS:
Drug: carboplatin — Given IV
Drug: cediranib maleate — Given orally
  Arms: Arm I
Drug: paclitaxel — Given IV
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving paclitaxel and carboplatin together with AZD2171 may kill more tumor cells. It is not yet known whether giving paclitaxel and carboplatin together with AZD2171 is more effective than giving paclitaxel and carboplatin together with a placebo in treating non-small cell lung cancer.

PURPOSE: This randomized phase II/III trial is studying how well giving paclitaxel and carboplatin together with cediranib maleate works and compares it to giving paclitaxel and carboplatin together with placebo in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival of patients with stage IIIB or IV non-small cell lung cancer treated with paclitaxel and carboplatin in combination with either cediranib maleate or a placebo.
* Determine the pharmacogenomics and pharmacodynamic aspects of these regimens in these patients. (Phase II)
* Compare the overall survival of patients treated with these regimens. (Phase III)

Secondary

* Compare objective tumor response rates in patients treated with these regimens.
* Determine the time to response and response duration in patients treated with these regimens. (Phase III)
* Determine the nature, severity, and frequency of the toxic effects of these regimens, including hemorrhage and hemoptysis, in these patients.
* Correlate the expression of tissue markers (at diagnosis) with outcomes and response in patients treated with these regimens. (Phase III)
* Compare quality of life of patients treated with these regimens. (Phase III)

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to gender, participating center, disease stage (IIIB vs IV), weight loss (≥ 5% vs < 5%), and prior adjuvant chemotherapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral cediranib maleate once daily in the absence of disease progression or unacceptable toxicity. Patients also receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment with paclitaxel and carboplatin repeats every 21 days for 6-8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive oral placebo once daily in the absence of disease progression or unacceptable toxicity. Patients also receive paclitaxel and carboplatin as in arm I.

Quality of life is assessed at baseline, before each treatment course, after completion of study treatment, and every 3 months thereafter.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 750 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), meeting 1 of the following stage criteria:

  * Stage IIIB disease

    * Patients without pleural effusion who are not candidates for combined modality treatment OR who were treated at centers where combined modality treatment is not considered standard treatment are eligible
  * Stage IV disease
* Measurable disease (phase II)

  * Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by x-ray, ultrasound, physical exam, or conventional CT scan OR ≥ 10 mm by spiral CT scan
  * Measurable lesions must be outside a previous radiotherapy field if they are the sole site of disease, unless disease progression has been documented
  * No significant central thoracic lesion with any appreciable cavitation
* Measurable or nonmeasurable disease (phase III)
* No necrotic or hemorrhagic tumor or metastases
* No untreated brain or meningeal metastases

  * CT scans are not required to rule out disease unless there is clinical suspicion of CNS disease
  * Patients with previously treated stable brain metastases (by radiography or clinical exam) are eligible provided they are asymptomatic and do not require corticosteroids

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No overt bleeding (i.e., ≥ 30 mL/episode) within the past 3 months

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2 times ULN (< 5 times ULN if liver metastases are present)

Renal

* Creatinine clearance ≥ 50 mL/min
* Proteinuria ≤ grade 1

Cardiovascular

* Mean QTc ≤ 470 msec (with Bazett's correction) by ECG
* No unstable angina
* No congestive heart failure
* No myocardial infarction within the past year
* No cardiac ventricular arrhythmias requiring medication
* No history of 2nd- or 3rd-degree atrioventricular conduction defects
* No untreated or uncontrolled cardiovascular condition
* No symptomatic cardiac dysfunction
* No uncontrolled hypertension (i.e., resting blood pressure ≥ 150/100 mm Hg despite antihypertensive therapy)
* No history of labile hypertension
* No history of poor compliance with antihypertensive medication
* No history of familial long-QT syndrome

Pulmonary

* No clinically relevant hemoptysis (i.e., ≥ 5 mL fresh blood) within the past 4 weeks

  * Flecks of blood only in sputum allowed

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective (double method for females; barrier method for males) contraception
* Able and willing to participate in the quality of life assessment
* No peripheral neuropathy > grade 1
* No prior allergic reaction to drugs containing Cremophor EL®
* No active or uncontrolled infection
* No serious illness or medical condition which would preclude study compliance
* No inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer or in situ cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 14 days since prior epidermal growth factor receptor-inhibitor therapy (e.g., tyrosine kinase inhibitor, monoclonal antibodies, vaccines, or other agents)
* No prior antiangiogenesis therapy, including any of the following:

  * Bevacizumab
  * Cediranib maleate
  * AZD6474
  * PTK787/ZK222584 (PTK/ZK)
  * Sunitinib malate
* Concurrent epoetin alfa allowed

Chemotherapy

* At least 12 months since prior adjuvant chemotherapy

  * Combined chemotherapy and radiotherapy regimens for locally advanced stage IIIB disease is not considered adjuvant therapy and is not allowed
* No prior chemotherapy for metastatic or recurrent NSCLC

Endocrine therapy

* See Disease Characteristics
* At least 1 week since prior steroids

Radiotherapy

* See Disease Characteristics
* At least 21 days since prior radiotherapy except for low-dose non-myelosuppressive radiotherapy with approval
* Concurrent palliative radiotherapy allowed with approval

Surgery

* At least 14 days since prior major surgery

Other

* Recovered from prior therapy
* Prior treatment with cyclooxygenase-2 inhibitors allowed
* Concurrent prophylactic anticoagulation (e.g., warfarin) allowed provided requirements for INR are met
* No potent inhibitors of CYP3A4 and 2C8, including any of the following drugs:

  * Amiodarone hydrochloride
  * Clarithromycin
  * Citalopram hydrobromide
  * Erythromycin
  * Omeprazole
  * Simvastatin
  * Atorvastatin
  * Lovastatin
  * Montelukast sodium
  * Verapamil hydrochloride
  * Ketoconazole
  * Miconazole
  * Indinovir and other antivrails
  * Diltiazem
* No other concurrent experimental drug or anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2005-11-03 (Actual); Primary Completion 2008-07-04 (Actual); Study Completion 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Toxicity | 3 years
Quality of Life | 3 years
Overall survival | 3 years
Correlative Studies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Glenwood D. Goss, MD, BCh, FCP, FRCPC, Study Chair — Ottawa Regional Cancer Centre; Scott A. Laurie, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre
Locations (20):
- Argentina (3):
  - Instituto Alexander Fleming, Buenos Aires
  - Compleso Medico de la Policia Federal Argentina, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
- Alfred Hospital, Melbourne, Australia
- Instituto Nacional de Cancer (INCA), Rio de Janeiro, Brazil
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Algoma District Cancer Program, Sault Ste. Marie, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - University Institute of Cardiology and, Québec, Quebec
- Romania (3):
  - Oncology Institute Bucharest, Bucharest
  - Oncological Institute "Ion Chiricuta", Cluj-Napoca
  - Clinical County Hospital of Sibiu, Sibiu
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradbury PA, Twumasi-Ankrah P, Ding K, et al.: The impact of brain metastases on overall survival (OS) in National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) clinical trials (CT) in advanced non-small cell lung cancer (NSCLC). [Abstract] J Clin Oncol 27 (Suppl 15): A-8075, 2009.
- [Result] Laurie SA, Gauthier I, Arnold A, Shepherd FA, Ellis PM, Chen E, Goss G, Powers J, Walsh W, Tu D, Robertson J, Puchalski TA, Seymour L. Phase I and pharmacokinetic study of daily oral AZD2171, an inhibitor of vascular endothelial growth factor tyrosine kinases, in combination with carboplatin and paclitaxel in patients with advanced non-small-cell lung cancer: the National Cancer Institute of Canada clinical trials group. J Clin Oncol. 2008 Apr 10;26(11):1871-8. doi: 10.1200/JCO.2007.14.4741. PMID 18398152
- [Result] Goss GD, Arnold A, Shepherd FA, Dediu M, Ciuleanu TE, Fenton D, Zukin M, Walde D, Laberge F, Vincent MD, Ellis PM, Laurie SA, Ding K, Frymire E, Gauthier I, Leighl NB, Ho C, Noble J, Lee CW, Seymour L. Randomized, double-blind trial of carboplatin and paclitaxel with either daily oral cediranib or placebo in advanced non-small-cell lung cancer: NCIC clinical trials group BR24 study. J Clin Oncol. 2010 Jan 1;28(1):49-55. doi: 10.1200/JCO.2009.22.9427. Epub 2009 Nov 16. PMID 19917841